CLINICAL TRIAL: NCT04075721
Title: A Phase I Open Label First in Human Dose Escalation of the Immunoproteasome Inhibitor M3258 as a Single Agent and Expansion Study of M3258 in Combination With Dexamethasone in Participants With Relapsed Refractory Multiple Myeloma
Brief Title: First in Human Dose Escalation of M3258 as a Single Agent and Expansion Study of M3258 in Combination With Dexamethasone
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was early discontinued due to lack of participant enrollment.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201814_0010; 2019-000947-28 (EudraCT Number)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: M3258; Dexamethasone; Pharmacokinetics; Relapsed Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — M3258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- M3258 10 mg QD (Experimental)
  Interventions: Drug: M3258
- M3258 10 mg Twice per Week (Experimental)
  Interventions: Drug: M3258
- M3258 20 mg Twice per Week (Experimental)
  Interventions: Drug: M3258 20 mg

INTERVENTIONS:
Drug: M3258 — Participants received M3258 at a dose of 10 milligrams (mg) orally, once daily (QD) or twice per week on Day 1 and Day 4 until disease progression.
  Arms: M3258 10 mg QD; M3258 10 mg Twice per Week
Drug: M3258 20 mg — Participants received M3258 at a dose of 20 mg orally, twice per week on Day 1 and Day 4 until disease progression.
  Arms: M3258 20 mg Twice per Week

SUMMARY:
The purpose of this study was to determine the safety, tolerability, pharmacokinetics, pharmacodynamics and early efficacy signs of M3258 as a single agent and co-administered with dexamethasone in participants with Relapsed Refractory Multiple Myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Participants having Eastern Co-operative Oncology Group (ECOG) Performance Status less than or equals to (<=) 1
* Adequate hematological, hepatic and renal function as defined in the protocol
* Participant must have measurable disease of Multiple Myeloma (MM) and received greater than (>) 3 prior lines of therapy for MM including a Proteasome Inhibitors (PI), an Immunomodulatory Imide Drug (IMiD) and an anti-CD38 mAb or who are refractory to at least PI agent (carfilzomib or bortezomib) and IMiD according to the International Myeloma Working Group (IMWG) criteria
* Participant must have documented evidence progressive disease as defined by the IMWG criteria either on or after their last regimen
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any condition, including any uncontrolled disease state that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
* An active second malignancy or evidence of disease of cancer (other than MM) before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence with the Sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
* Cerebrovascular accident/stroke (< 6 months prior enrollment) or neurologic instability per clinical evaluation due to tumor involvement of the Central Nervous System
* Diagnosis of fever within 1 week prior to study intervention administration
* Part B: Participants planning to undergo a stem cell transplant should not be enrolled to reduce disease burden prior to transplant.
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (7):
- United States (4):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Georgetown University Medical Center- Research Parent, Washington D.C., District of Columbia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Sarah Cannon Research Institute, Nashville, Tennessee
- France (3):
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Vauvert

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- [Result] Sanderson MP, Friese-Hamim M, Walter-Bausch G, Busch M, Gaus S, Musil D, Rohdich F, Zanelli U, Downey-Kopyscinski SL, Mitsiades CS, Schadt O, Klein M, Esdar C. M3258 Is a Selective Inhibitor of the Immunoproteasome Subunit LMP7 (beta5i) Delivering Efficacy in Multiple Myeloma Models. Mol Cancer Ther. 2021 Aug;20(8):1378-1387. doi: 10.1158/1535-7163.MCT-21-0005. Epub 2021 May 27. PMID 34045234
- [Derived] Lignet F, Esdar C, Walter-Bausch G, Friese-Hamim M, Stinchi S, Drouin E, El Bawab S, Becker AD, Gimmi C, Sanderson MP, Rohdich F. Translational PK/PD Modeling of Tumor Growth Inhibition and Target Inhibition to Support Dose Range Selection of the LMP7 Inhibitor M3258 in Relapsed/Refractory Multiple Myeloma. J Pharmacol Exp Ther. 2023 Jan;384(1):163-172. doi: 10.1124/jpet.122.001355. Epub 2022 Oct 23. PMID 36273822
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201814_0010
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent: 26 September 2019, Last participant last visit: 01 April 2021.
Pre-assignment Details: This study was planned to be conducted in 2 parts; Part A: Dose escalation part and Part B: Dose expansion part. However, because of early discontinuation, only Part A was conducted; due to lack of participant enrollment before Part A reached its primary objective and before Part B was started.
Groups:
- M3258 10 mg QD: Participants received M3258 at a dose of 10 milligrams (mg) orally, once daily (QD) until disease progression.
- M3258 10 mg Twice Per Week: Participants received M3258 at a dose of 10 mg orally, twice per week on Day 1 and Day 4 until disease progression.
- M3258 20 mg Twice Per Week: Participants received M3258 at a dose of 20 mg orally, twice per week on Day 1 and Day 4 until disease progression.
Period: Overall Study
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Started | 2 | 4 | 4
Pharmacokinetic (PK) Analysis Set | 2 | 5 (1 participant received actual dose of 10 mg in Cycle 1 Day 1 instead of planned 20 mg and was summarized with the 10 mg dose level for PK analysis set.) | 3
Pharmacodynamics (Pd) Analysis Set | 2 | 5 (1 participant received actual dose of 10 mg in Cycle 1 Day 1 instead of planned 20 mg and was summarized with the 10 mg dose level for Pd analysis set.) | 3
Completed | 2 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week | Total
Number analyzed (Participants) | 2 | 4 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 4
  >=65 years | 1 | 2 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 4 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 0 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-Limiting Toxicities (DLTs) as Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: DLT: any of adverse events (AEs), assessed by Investigator and/Sponsor at any dose, regimen, and judged not to be related to underlying disease/any previous/concomitant medication/concurrent condition during first cycle of study treatment. DLT was confirmed by Safety Monitoring Committee. DLTs: Grade (Gr) greater than/equal to (>=) 3 nonhematologic AE with exception of: Single laboratory values out of abnormal range; Gr3 diarrhea persisting less than or equal to [<=] 72 hour (hr); Nausea and vomiting <= 72 hr; Transient Gr3 fatigue, local reactions, flu-like symptoms <= 72 hr; Gr3 nonrecurrent skin toxicity; Asymptomatic Gr >= 3 lipase/amylase elevation. Any Gr >= 4 hematologic AE: Gr >= 3 febrile neutropenia with Absolute Neutrophil Count (ANC) <1000 per cube millimeter and temperature of >38.3 Celsius (°C); Gr >= 3 thrombocytopenia; Gr4 thrombocytopenia lasting >7 days.
Time Frame: Day 1 up to Day 28
Population: DLT analysis set: all participants who received at least 1 dose of study intervention and meet at least 1 of criteria specified in statistical analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 3
Participants | 1 | 0 | 1

2. Primary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Event (TEAEs) and Treatment-Related Adverse Event (TRAEs)
Description: Adverse Event (AE): any untoward medical occurrence in a participant administered with a study drug, which does not necessarily have a causal relationship with this treatment. TEAEs: events that started from first dose of study intervention to 30 days after end of study intervention, or the cutoff date, whichever occurred first. TEAEs included both serious TEAEs (Serious AE: AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect) and non-serious TEAEs. TRAEs are defined as those AEs which are reasonably related to the study intervention.
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Participants with TEAEs | 2 | 4 | 4
  Participants with TRAEs | 2 | 3 | 3

3. Primary Outcome: Part A: Number of Participants With Treatment-Emergent Adverse Event (TEAEs) Outside of Dose-Limiting Toxicity (DLT) Period That Safety Monitoring Committee Deems Relevant for Determination of the Maximum Tolerated Dose
Description: as for outcome 2
Time Frame: Day 29 up to 20.1 weeks
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants | 0 | 0 | 0

4. Primary Outcome: Part A: Change From Baseline in 12-lead Electrocardiogram (ECG) Findings: QT Interval - Fridericia's Correction Formula
Description: 12-lead ECG were recorded after the participants have rested for at least 15 minutes in supine position. Change from baseline in 12-Lead ECG findings that is QT interval - Fridericia's correction formula at pre-dose on Cycle 2 Day 1 were reported.
Time Frame: Cycle 1 Day 1 pre-dose (Baseline), pre-dose on Cycle 2 Day 1 (each Cycle is of 28 days)
Population: Safety analysis set included all participants who were administered any dose of the study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: milliseconds (msec)
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 1 | 3 | 1
milliseconds (msec) | -10.0 (-10) [-10 to -10] | 6.3 (-17) [-17 to 45] | 6.0 (6) [6 to 6]

5. Primary Outcome: Part A: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: ECOG performance status measured to assess participant's performance status on a scale of 0 to 5, where 0 = Fully active, able to carry on all pre-disease activities without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; 3 = Capable of only limited self-care, confined to bed/chair for more than 50 percent of waking hours; 4 = Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5 = dead. ECOG performance status was reported in terms of number of participants with shifts in score from baseline value vs worst post-baseline value (that is [i.e.] highest score).
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Baseline score 0, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 1 | 1 | 2 | 1
  Baseline score 0, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 3 | 0 | 0 | 1
  Baseline score 0, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 0, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 0 | 1 | 1 | 0
  Baseline score 1, worst post-baseline score 1 | 0 | 1 | 0
  Baseline score 1, worst post-baseline score 2 | 0 | 0 | 1
  Baseline score 1, worst post-baseline score 3 | 0 | 0 | 1
  Baseline score 1, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 1, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 1 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 3 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 2, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 1 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 3 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 3, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 1 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 3 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 4, worst post-baseline score 5 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 0 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 1 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 2 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 3 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 4 | 0 | 0 | 0
  Baseline score 5, worst post-baseline score 5 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Shift From Baseline Grade Less Than (<) 3 in Clinical Laboratory Parameters to Grade Greater Than or Equal to (>=) 3 on Treatment
Description: Laboratory parameters included hematology, chemistry, and coagulation. Number of participants with shifts from baseline (Grade <3) to >= Grade 3 were reported as per NCI-CTCAE, v5.0 graded from Grade 1 to 5. Grade 1: Mild, Grade 2: Moderate; Grade 3: Severe. Grade 4: Life-threatening and Grade 5: Death.
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Hematology | 2 | 3 | 4
  Chemistry | 0 | 0 | 3
  Coagulation | 0 | 0 | 0

7. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Changes From Baseline in Vital Signs - Maximal Body Temperature Increase
Description: The number of participants with treatment-emergent changes from baseline in increased Body Temperature (degree Celsius [°C]) were reported by using criteria: Baseline temperature (temp.) less than (<) 37°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C and greater than or equal to (>=)3°C; Baseline temp. 37 - <38°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C and >=3°C; Baseline temp. 38 - <39°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C and >=3°C; Baseline temp. 39-<40°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C and >=3°C; Baseline temp. >=40°C, on treatment change <1°C, 1 - <2°C, 2 - <3°C and >=3°C.
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Baseline temp. <37°C, on treatment change <1°C | 0 | 1 | 2
  Baseline temp.<37°C, on treatment change 1 - <2°C | 2 | 0 | 1
  Baseline temp. <37°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. <37°C, on treatment change >=3°C | 0 | 1 | 0
  Baseline temp. 37 - <38°C, on treatment change <1°C | 0 | 2 | 1
  Baseline temp. 37 - <38°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. 37 - <38°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 37 - <38°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change <1°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 38 - <39°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change <1°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. 39 - <40°C, on treatment change >=3°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change <1°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change 1 - <2°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change 2 - <3°C | 0 | 0 | 0
  Baseline temp. >=40°C, on treatment change >=3°C | 0 | 0 | 0

8. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Changes From Baseline in Vital Signs - Maximal Systolic Blood Pressure Increase/Decrease and Maximal Diastolic Blood Pressure Increase/Decrease
Description: The number of participants with treatment-emergent changes from baseline (BS) in Increase (Ic.)/Decrease (Dc.) Systolic Blood Pressure (SBP) and diastolic blood pressure (DBP) (millimeter of mercury [mmHg]) were reported by using criteria: Ic./Dc. BS SBP/DBP <140/<90 mmHg, on maximal treatment (TR) change =<20 mmHg, >20 - =<40 mmHg and >40 mmHg; Ic./Dc. BS SBP/DBP >=140/>=90 mmHg, on maximal TR change =<20 mmHg, >20 - =<40 mmHg and >40 mmHg.
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Ic. BS SBP <140 mmHg, on TR change =<20 mmHg | 0 | 1 | 1
  Ic. BS SBP <140 mmHg, on TR change >20 - =<40 mmHg | 1 | 1 | 1
  Ic. BS SBP <140 mmHg, on TR change >40 mmHg | 1 | 1 | 1
  Ic. BS SBP >=140 mmHg, on TR change =<20 mmHg | 0 | 1 | 1
  Ic. BS SBP >=140 mmHg, on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Ic. BS SBP >=140 mmHg, on TR change >40 mmHg | 0 | 0 | 0
  Dc. BS SBP <140 mmHg, on TR change =<20 mmHg | 2 | 3 | 3
  Dc. BS SBP <140 mmHg, on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Dc. BS SBP <140 mmHg, on TR change >40 mmHg | 0 | 0 | 0
  Dc. BS SBP >=140 mmHg, on TR change =<20 mmHg | 0 | 1 | 1
  Dc. BS SBP >=140 mmHg, on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Dc. BS SBP >=140 mmHg, on TR change >40 mmHg | 0 | 0 | 0
  Ic. BS DBP <90 mmHg, on TR change =<20 mmHg | 1 | 1 | 3
  Ic. BS DBP <90 mmHg, on TR change >20 - =<40 mmHg | 1 | 1 | 0
  Ic. BS DBP <90 mmHg, on TR change >40 mmHg | 0 | 1 | 0
  Ic. BS DBP >=90 mmHg, on TR change =<20 mmHg | 0 | 1 | 1
  Ic. BS DBP >=90 mmHg, on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Ic. BS DBP >=90 mmHg, on TR change >40 mmHg | 0 | 0 | 0
  Dc. BS DBP <90 mmHg, on TR change =<20 mmHg | 2 | 3 | 3
  Dc. BS DBP <90 mmHg, on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Dc. BS DBP <90 mmHg, on TR change >40 mmHg | 0 | 0 | 0
  Dc. BS DBP >=90 mmHg, on TR change =<20 mmHg | 0 | 1 | 1
  Dc. BS DBP >=90 mmHg,on TR change >20 - =<40 mmHg | 0 | 0 | 0
  Dc. BS DBP >=90 mmHg, on TR change >40 mmHg | 0 | 0 | 0

9. Secondary Outcome: Part A: Number of Participants With Treatment-Emergent Changes From Baseline in Vital Signs - Maximal Respiration Rate Increase/Decrease
Description: The number of participants with treatment-emergent changes from baseline in Increase (Ic.)/Decrease (Dc.) maximal Respiration Rate (RR) were reported by using criteria: Ic./Dc. BS RR <20 breaths per minute (breaths/min), on TR change (ch) =<5 breaths/min, >5 - =<10 breaths/min and >10 breaths/min. Ic./Dc. BS RR >=20 breaths/min, on TR ch =<5 breaths/min, >5 - =<10 breaths/min and >10 breaths/min.
Time Frame: Time from first treatment up to 30 days after end of study intervention (assessed up to 24.3 weeks)
Population: Safety analysis set included all participants who were administered any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Ic. BS RR <20 breaths/min, on TR ch =<5 breaths/min | 2 | 1 | 2
  Ic.BS RR<20 breaths/min, on TR Ch >5 - = <10 breaths/min | 0 | 1 | 2
  Ic. BS RR <20 breaths/min, on TR ch >10 breaths/min | 0 | 0 | 0
  Ic. BS RR >=20 breaths/min, on TR ch =<5 breaths/min | 0 | 2 | 0
  IC.BS RR >=20 breaths/min, on TR ch >5 - =<10 breaths/min | 0 | 0 | 0
  Ic. BS RR >=20 breaths/min, on TR ch >10 breaths/min | 0 | 0 | 0
  Dc. BS RR <20 breaths/min, on TR ch =<5 breaths/min | 2 | 2 | 4
  Dc. BS RR <20 breaths/min, on TR Ch >5 - =<10 breaths/min | 0 | 0 | 0
  Dc. BS RR <20 breaths/min, on TR ch >10 breaths/min | 0 | 0 | 0
  Dc. BS RR >=20 breaths/min, on TR ch =<5 breaths/min | 0 | 2 | 0
  Dc.BS RR >=20 breaths/min, on TR ch >5 - =<10 breaths/min | 0 | 0 | 0
  Dc. BS RR >=20 breaths/min, on TR ch >10 breaths/min | 0 | 0 | 0

10. Secondary Outcome: Part A: Single Dose: Maximum Observed Plasma Concentration (Cmax) of M3258
Description: Cmax was obtained directly from the concentration versus time curve. Single dose PK data on Day 1 were summarized by dose level, such that all 10 mg arms were combined as descriptive statistics of PK were only calculated for N greater than (>) 2 in which a measurement of greater than (>) lower limit of quantification (LLOQ) represents a valid measurement.
Time Frame: Cycle 1 Day 1: Pre-dose 1, 2, 3, 4, 5, 6, 8 and 24 hours post-dose (each Cycle is of 28 days)
Population: Pharmacokinetic (PK) analysis set included all participants, who received at least one dose of study intervention, have no clinically important protocol deviations or important events affecting PK, and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Groups:
- M3258 10 mg QD or Twice Per Week: Participants received M3258 at a dose of 10 mg orally, QD or twice per week until disease progression.
Arm/Group | M3258 10 mg QD or Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 5 | 3
nanogram per milliliter (ng/mL) | 153 [151 to 156] | 215 [206 to 223]

11. Secondary Outcome: Part A: Mutilple Dose: Maximum Observed Plasma Concentration (Cmax) of M3258
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Cycle 1 Day 8 or Cycle 1 Day 15: Pre-dose 1, 2, 3, 4, 5, 6, and 8 hours post-dose (each Cycle is of 28 days)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Groups:
- M3258 10 mg Twice Per Week: Participants received M3258 at a dose of 10 mg orally, twice per week until disease progression.
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 1 | 3 | 3
nanogram per milliliter (ng/mL) | NA [NA to NA] — Based on pre-specified criteria Geometric Mean and 95% Confidence Interval were not calculated if fewer than 2 participants have reportable parameter values. | 213 [208 to 217] | 511 [507 to 516]

12. Secondary Outcome: Part A: Single Dose: Area Under Plasma Concentration-Time Curve (AUC) From Time Zero to Last Sampling Time (AUC0-t) of M3258
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule. Single dose PK data on Day 1 were summarized by dose level, such that all 10 mg arms were combined as descriptive statistics of PK were only calculated for N greater than (>) 2 in which a measurement of greater than (>) lower limit of quantification (LLOQ) represents a valid measurement.
Time Frame: Cycle 1 Day 1: Pre-dose 1, 2, 3, 4, 5, 6, 8 and 24 hours post-dose (each Cycle is of 28 days)
Population: PK analysis set included all participants, who received at least one dose of study intervention, have no clinically important protocol deviations or important events affecting PK, and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | M3258 10 mg QD or Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 5 | 3
hour*nanogram per milliliter (h*ng/mL) | 2000 [2000 to 2010] | 3300 [3300 to 3310]

13. Secondary Outcome: Part A: Single Dose: Area Under Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of M3258
Description: Area under the plasma concentration versus time curve from time zero to 24 hours post dosing for M3258. Single dose PK data on Day 1 were summarized by dose level, such that all 10 mg arms were combined as descriptive statistics of PK were only calculated for N greater than (>) 2 in which a measurement of greater than (>) lower limit of quantification (LLOQ) represents a valid measurement.
Time Frame: Cycle 1 Day 1: Pre-dose 1, 2, 3, 4, 5, 6, 8 and 24 hours post-dose (each Cycle is of 28 days)
Population: The most participants who had evaluable PK, samples at 24 hour (Day 2) were collected. Therefore, the AUC0-t and AUC0-24 would not differ and AUC0-24 at single dose was not reported. It was also planned to carry the trough value at steady state for QD dosing forward and impute it as trough value at 24 hours. Due to the change from the QD to twice per week dosing this did not apply anymore and AUC0-24 at steady state was not calculated.
Arm/Group | M3258 10 mg QD or Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part A: Multiple Dose: Area Under Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of M3258
Description: Area under the plasma concentration versus time curve from time zero to 24 hours post dosing for M3258.
Time Frame: Cycle 1 Day 8 or Cycle 1 Day 15: Pre-dose 1, 2, 3, 4, 5, 6, and 8 hours post-dose (each Cycle is of 28 days)
Population: as for outcome 13
Arm/Group | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week | M3258 10 mg QD
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Part A: Single Dose: Ratio to Baseline in Large Multifunctional Protease 7 (LMP7) Activity at Cycle 1 Day 1
Description: Ratio to baseline was calculated dividing post-baseline measurements by the baseline measurement. Single dose Pd data on Day 1 were summarized by dose level, such that all 10 mg arms were combined as descriptive statistics of PK were only calculated for N greater than (>) 2 in which a measurement of greater than (>) lower limit of quantification (LLOQ) represents a valid measurement.
Time Frame: Baseline (Pre-dose), 2, 6 and 24 hours post-dose on Cycle 1 Day 1 (each Cycle is of 28 days)
Population: The Pharmacodynamic (Pd) population included all participants who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting Pd, and provide at least one measurable Pd endpoint post-dose. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified timepoints.
Measure: Mean (Full Range); unit: ratio
Arm/Group | M3258 10 mg QD or Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 3 | 2
ratio
  Cycle 1 Day 1: 2 hours post-dose | 0.308 [0.21 to 0.41] | 0.370 [0.31 to 0.43]
  Cycle 1 Day 1: 6 hours post-dose | 0.337 [0.20 to 0.55] | 0.178 [0.15 to 0.21]
  Cycle 1 Day 1: 24 hours post-dose: number analyzed (Participants) | 2 | 2
  Cycle 1 Day 1: 24 hours post-dose | 0.387 [0.25 to 0.53] | 0.262 [0.16 to 0.36]

16. Secondary Outcome: Part A: Multiple Dose: Ratio to Baseline in Large Multifunctional Protease 7 (LMP7) Activity at Cycle 1 Day 8 (or Day 15)
Description: Ratio to baseline was calculated dividing post-baseline measurements by the baseline measurement.
Time Frame: Cycle 1 Day 1 pre-dose (Baseline), Pre-dose, 2 and 6 hours post-dose on Cycle 1 Day 8 (or Day 15) (each Cycle is of 28 days)
Population: The Pd population included all participants who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting Pd, and provide at least one measurable Pd endpoint post-dose. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified timepoints.
Measure: Mean (Full Range); unit: ratio
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 1 | 2 | 2
ratio
  Cycle 1 Day 8 (or Day 15): Pre-dose: number analyzed (Participants) | 1 | 2 | 1
  Cycle 1 Day 8 (or Day 15): Pre-dose | 0.26 [0.26 to 0.26] | 0.364 [0.36 to 0.37] | 0.31 [0.31 to 0.31]
  Cycle 1 Day 8 (or Day 15): 2 hours post-dose | 0.25 [0.25 to 0.25] | 0.202 [0.17 to 0.24] | 0.299 [0.16 to 0.44]
  Cycle 1 Day 8 (or Day 15): 6 hours post-dose: number analyzed (Participants) | 0 | 2 | 1
  Cycle 1 Day 8 (or Day 15): 6 hours post-dose |  | 0.178 [0.17 to 0.19] | 0.22 [0.22 to 0.22]

17. Secondary Outcome: Part A: Change From Baseline in Serum Monoclonal (M)-Protein Level Measured Using Electrophoresis
Description: Change from baseline in serum monoclonal (M)-protein level was measured by using electrophoresis at Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and end of study intervention.
Time Frame: Baseline, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and end of study intervention (Week 20.1) (each Cycle is of 28 days)
Population: Safety analysis set included all participants who were administered any dose of the trial medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified timepoints.
Measure: Mean (Full Range); unit: gram per deciliter (g/dL)
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 1 | 4 | 3
gram per deciliter (g/dL)
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 3 | 1
  Cycle 2 Day 1 |  | -0.113 [-0.21 to -0.05] | 0.000 [0.00 to 0.00]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 3 | 1
  Cycle 3 Day 1 |  | 0.107 [-0.14 to 0.36] | 0.100 [0.10 to 0.10]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 3 | 0
  Cycle 4 Day 1 |  | 0.050 [-0.08 to 0.23] |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 6 Day 1 |  | 0.100 [0.10 to 0.10] |
  End of Study Intervention | 0.100 [0.10 to 0.10] | 0.678 [0.27 to 1.68] | 1.223 [0.68 to 1.91]

18. Secondary Outcome: Part A: Change From Baseline in Urine M-protein Level Using Electrophoresis
Description: Change from baseline in urine M-protein level was measured by using electrophoresis at Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and end of study intervention.
Time Frame: as for outcome 17
Population: Safety analysis set included all participants who were administered any dose of the trial medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified timepoints. None of the participants were analyzed in M3258 10 mg QD arm at specified timepoints.
Measure: Mean (Full Range); unit: milligrams per day (mg/day)
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 0 | 2 | 1
milligrams per day (mg/day)
  Cycle 2 Day 1 |  | 25.25 [-59.5 to 110.0] | 26.50 [26.5 to 26.5]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 3 Day 1 |  | 256.00 [256.0 to 256.0] | 67.00 [67.0 to 67.0]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 4 Day 1 |  | -130.00 [-130.0 to 130.0] |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 5 Day 1 |  | 268.00 [268.0 to 268.0] |
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 6 Day 1 |  | 3320.00 [3320.0 to 3320.0] |
  End of Study Intervention: number analyzed (Participants) | 0 | 2 | 0
  End of Study Intervention |  | 610.50 [51.0 to 1170.0] |

19. Secondary Outcome: Part A: Change From Baseline in Free Light Chain Ratio
Description: Change from baseline in free light chain ratio was reported at Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1 and end of study intervention.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Full Range); unit: ratio
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 1 | 1
ratio
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 1
  Cycle 2 Day 1 | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 3 Day 1 |  | 0.000 [0.00 to 0.00] | 0.010 [0.01 to 0.01]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 4 Day 1 |  | 0.000 [0.00 to 0.00] |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 5 Day 1 |  | 0.000 [0.00 to 0.00] |
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Cycle 6 Day 1 |  | -0.010 [-0.01 to -0.01] |
  End of Study Intervention | -0.005 [-0.01 to 0.00] | -0.010 [-0.01 to -0.01] | 0.000 [0.00 to 0.00]

20. Secondary Outcome: Part A: Number of Participants With Overall Response (OR) as Assessed by Investigator Using International Myeloma Working Group (IMWG) Criteria
Description: OR is defined as a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) based on the IMWG Criteria: sCR: CR (negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow); normal free light chain (FLC) ratio and no clonal cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis/>= 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: >= 50% reduction of serum M-Protein and reduction in urinary M-protein by >= 90%/to < 200 mg/24 hours. In addition to the above, if present at baseline a >= 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Time from first dose of study treatment up to 18.2 months
Population: Safety analysis set included all participants who were administered any dose of the trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Stringent Complete Response | 0 | 0 | 0
  Complete Response | 0 | 0 | 0
  Very good Partial Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0

21. Secondary Outcome: Duration of Response (DoR) as Assessed by Investigator Using International Myeloma Working Group (IMWG) Criteria
Description: DOR was defined participants with confirmed response, as time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to date of first documentation of progression disease (PD)/death due to any cause, whichever occurred first. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. PR: >= 50% reduction of serum M-Protein and reduction in urinary M-protein by >= 90%/to < 200 mg/24 hours. In addition to the above, if present at baseline a >= 50% reduction in the size of soft tissue plasmacytomas is also required. PD: >= 25% increase from lowest response value in serum. Development of new or increased size of existing bone lesions or soft tissue plasmacytomas. Hypercalcemia attributed to the plasma cell proliferative disorder.
Time Frame: Time from first documentation of objective response until date of first documentation of PD or death due to any cause, whichever occurred first, assessed up to 18.2 months
Population: Data could not be calculated as none of the participants showed objective response.
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Time to Response as Assessed by Investigator Using International Myeloma Working Group (IMWG) Criteria
Description: Time to response was defined as the time from the first dose of M3258 to the documentation of first response (Complete Response [CR] or Partial Response [PR]). CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. PR: >= 50% reduction of serum M-Protein and reduction in urinary M-protein by >= 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a >= 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Time from the first dose of study treatment up to documentation of first response, assessed up to 18.2 months
Population: Data could not be calculated as none of the participants showed response.
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from first treatment up to final assessment at 18.2 months
Description: Safety analysis set included all participants who were administered any dose of the study medication.
Arm/Group | M3258 10 mg QD | M3258 10 mg Twice Per Week | M3258 20 mg Twice Per Week
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 3/4 | 3/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M3258 10 mg QD (N=2) | M3258 10 mg Twice Per Week (N=4) | M3258 20 mg Twice Per Week (N=4)
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Spinal cord haemorrhage (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M3258 10 mg QD (N=2) | M3258 10 mg Twice Per Week (N=4) | M3258 20 mg Twice Per Week (N=4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Part B was not conducted as the study was early discontinued due to lack of participant's recruitment into Part A before Part A reached its primary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04075721/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04075721/SAP_001.pdf